CLINICAL TRIAL: NCT00609193
Title: Functional and Neurochemical Brain Changes in First-episode Bipolar Mania Following Successful Treatment With Lithium or Quetiapine
Brief Title: Functional and Neurochemical Brain Changes in First-episode Bipolar Mania
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Stephen Strakowski, Academic Director of Medicine, University of Cincinnati
Other Study IDs: BITREC - Project I
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Quetiapine Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Study subjects receiving lithium
  Interventions: Drug: lithium
- 2: Study subjects receiving quetiapine
  Interventions: Drug: quetiapine

INTERVENTIONS:
Drug: lithium — standard clinical care
  Groups: 1
Drug: quetiapine — standard clinical care
  Groups: 2

SUMMARY:
The purpose of this study is to use magnetic resonance imaging (MRI) to examine brain structure, function and chemistry in people with bipolar disorder who are being treated with either quetiapine or lithium. Both of these medicines are FDA-approved to treat mania in adults and lithium is also FDA approved in children; quetiapine is commonly used in children with mania, but is not FDA approved for this indication in this age group.

ELIGIBILITY:
Inclusion Criteria - First-episode manic bipolar patients (N=100; 15-20 patients/year):

1. Patients meet DSM-IV criteria for type I bipolar disorder, manic or mixed.
2. Patients have an index Young Mania Rating Scale (YMRS)70 total score >20.
3. Patients have <3 months of lifetime anti-manic or anti-depressant medication exposure, including no active psychotropic medication in the one weeks prior to the index admission. Importantly, patients will NOT be taken off medications for this study; this criterion is to exclude subjects receiving active treatment at the time of admission to support the 'first-episode' criterion.
4. Patients have no more than two prior episodes of major depression.
5. Patients are between 12 and 35 years old; subjects < 18 yrs old have a Tanner greater than or equal to 4

Exclusion criteria: All subjects will be excluded from participation for the following reasons.

1. Any chemical use disorder within 3 months.
2. Any medical or neurological disorder that could influence fMRI and MRS results.
3. A history of mental retardation or an estimated IQ total score <85.
4. An MRI scan is contraindicated in the subject.
5. The patient cannot attend follow-up visits.
6. A positive urine pregnancy test (in women).

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: You are being asked to take part in this research study because you have been diagnosed with bipolar disorder and are currently experiencing mania. Mania is identified by periods of extreme elation or irritability, excessive energy, racing thoughts, difficulty sleeping, poor judgment and/or reckless behavior. Bipolar disorder is an illness in which people experience mania as well as mood swings into depression. To participate in this study you must be at least 12 years old and no older than 35.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2008-01; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to use magnetic resonance imaging (MRI) to examine brain structure, function and chemistry in people with bipolar disorder who are being treated with either quetiapine or lithium. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Strakowski, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Lei D, Li W, Tallman MJ, Strakowski SM, DelBello MP, Rodrigo Patino L, Fleck DE, Lui S, Gong Q, Sweeney JA, Strawn JR, Nery FG, Welge JA, Rummelhoff E, Adler CM. Changes in the structural brain connectome over the course of a nonrandomized clinical trial for acute mania. Neuropsychopharmacology. 2022 Oct;47(11):1961-1968. doi: 10.1038/s41386-022-01328-y. Epub 2022 May 18. PMID 35585125
- [Derived] Lippard ETC, Weber W, Welge J, Adler CM, Fleck DE, Almeida J, DelBello MP, Strakowski SM. Variation in rostral anterior cingulate functional connectivity with amygdala and caudate during first manic episode distinguish bipolar young adults who do not remit following treatment. Bipolar Disord. 2021 Aug;23(5):500-508. doi: 10.1111/bdi.13025. Epub 2020 Nov 18. PMID 33089593
- [Derived] Strakowski SM, Fleck DE, Welge J, Eliassen JC, Norris M, Durling M, Komoroski RA, Chu WJ, Weber W, Dudley JA, Blom TJ, Stover A, Klein C, Strawn JR, DelBello MP, Lee JH, Adler CM. fMRI brain activation changes following treatment of a first bipolar manic episode. Bipolar Disord. 2016 Sep;18(6):490-501. doi: 10.1111/bdi.12426. Epub 2016 Sep 19. PMID 27647671